CLINICAL TRIAL: NCT02915367
Title: Next Generation Real-time Monitoring for PrEP Adherence in Young Kenyan Women
Brief Title: Monitoring Pre-exposure Prophylaxis for Young Adult Women
Acronym: MPYA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: University of Washington (Other); Kenya Medical Research Institute (Other)
Responsible Party: Principal Investigator, Jessica Haberer, MD, Research Scientist, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: R01MH109309 (NIH)
Record Dates: First submitted 2016-09-16; First posted 2016-09-27 (Estimated); Results first posted 2022-04-08 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-04

CONDITIONS: HIV/AIDS; Adherence
Keywords: HIV/AIDS; adherence; women; real time monitoring; risk; SMS; mHealth
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SMS Reminders (Experimental): Participants will receive regular SMS reminders regarding PrEP. All participants will receive adherence monitoring through a WisePill device.
  Interventions: Behavioral: SMS Reminders
- No Reminders (No Intervention): Participants will not receive SMS reminders. All participants will receive adherence monitoring through a WisePill device.

INTERVENTIONS:
Behavioral: SMS Reminders — Participants will receive daily reminders, with content and timing of their choosing, regarding their PrEP use. Participants will have the choice to later receive SMS reminders only when they forget to take their dose (as indicated by real-time adherence monitoring via WisePill).
  Arms: SMS Reminders

SUMMARY:
Next generation real-time monitoring for PrEP adherence in young Kenyan women

DETAILED DESCRIPTION:
This protocol describes a longitudinal study of young Kenyan women at high risk for HIV who will be offered HIV pre-exposure prophylaxis (PrEP) for up to two years. Adherence will be monitored in all women with the next generation Wisepill; half will be randomized to receive short message service (SMS) reminders. The technical function, acceptability, cost, and validity of the next generation Wisepill device coupled to SMS reminders will be determined among this cohort of young Kenyan women. Additionally, SMS will be used for longitudinal assessment of risk perception and its alignment with PrEP adherence.

ELIGIBILITY:
Inclusion Criteria:

* HIV-uninfected (as determined by Kenya national testing algorithms)
* Wanting to start PrEP with an initial recommendation of 6 months of use
* Clinically safe to receive PrEP, in accordance with Centers for Disease Control and Prevention (CDC) guidelines:

  * Creatinine clearance >60 mL/min
  * Not infected with hepatitis B
  * No other medical condition that in the discretion of the site investigator would make participation unsafe or complicate the goals of the study
* Sexually active (defined as vaginal or anal sex) within the last 3 months
* At high risk for HIV infection based on a validated risk score of >5 or being in an HIV serodiscordant relationship
* Not pregnant
* Owns a personal cell phone (not shared) compatible with study protocols and the ability to charge it
* Ability to send a text message
* Intending to stay in the area for at least the next year
* Willing to use study criteria

Exclusion Criteria:

* Unable to provide consent
* Breast-feeding (PrEPis not currently approved for use during breast-feeding)
* Concurrent participation in another research study that may influence adherence to PrEP and/or interfere with the procedures of this study.

Ages: 18 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 348 (Actual)
Dates: Start 2016-12-21 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2020-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Haberer, MD, MS, Principal Investigator — Massachussetts General Hospital; Jared Baeten, MD, PhD, Principal Investigator — University of Washington; Nelly Mugo, Study Director — Kenya Medical Research Institute; Elizabeth Bukusi, Study Director — Kenya Medical Research Institute
Locations (2):
- Kenya (2):
  - KEMRI, Kisumu
  - KEMRI, Thika

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be made available at the end of the study upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available within 12 months of publishing primary results
Access Criteria: Data use agreement

REFERENCES:
- [Derived] Haberer JE, Mugo N, Bukusi EA, Ngure K, Kiptinness C, Oware K, Garrison LE, Musinguzi N, Pyra M, Valenzuela S, Thomas KK, Anderson PL, Thirumurthy H, Baeten JM. Understanding Pre-Exposure Prophylaxis Adherence in Young Women in Kenya. J Acquir Immune Defic Syndr. 2022 Mar 1;89(3):251-260. doi: 10.1097/QAI.0000000000002876. PMID 35147580
- [Derived] Haberer JE, Bukusi EA, Mugo NR, Pyra M, Kiptinness C, Oware K, Garrison LE, Thomas KK, Musinguzi N, Morrison S, Anderson PL, Ngure K, Baeten JM; MPYA Study Team. Effect of SMS reminders on PrEP adherence in young Kenyan women (MPYA study): a randomised controlled trial. Lancet HIV. 2021 Mar;8(3):e130-e137. doi: 10.1016/S2352-3018(20)30307-6. PMID 33662265

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SMS Reminders | No Reminders
Started | 173 | 175
Completed | 136 | 144
Not Completed | 37 | 31

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SMS Reminders | No Reminders | Total
Number analyzed (Participants) | 173 | 175 | 348
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 15 | 19 | 34
  Between 18 and 65 years | 158 | 156 | 314
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 21 [19 to 22] | 21 [19 to 22] | 21 [19 to 22]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 173 | 175 | 348
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 173 | 175 | 348
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Kenya | 173 | 175 | 348

OUTCOME MEASURES:

1. Primary Outcome: Enacted Adherence as Measured by Electronic Monitoring at 6 and 24 Months
Description: Comparison of average percent adherence (doses taken/doses prescribed) by study arm at each time point among participants choosing to pick up PrEP.
Time Frame: up to 2 years follow-up
Population: Number of participants choosing to take PrEP per arm
Measure: Mean (95% Confidence Interval); unit: percentage of adherence
Arm/Group | SMS Reminders | No Reminders
Number analyzed (Participants) | 173 | 175
percentage of adherence
  Month 6 adherence | 40.2 [36.1 to 44.4] | 36.8 [32.7 to 40.8]
  Month 24 adherence | 27.0 [23.6 to 30.5] | 26.6 [23.1 to 30.2]

2. Secondary Outcome: Number of Participants Reporting High Acceptability of Wisepill Devices for PrEP Adherence Monitoring
Description: Questionnaire indicating "very interested" in using the Wisepill monitor (a pill box that records the date and time of each opening as a proxy for pill ingestion)
Time Frame: Month 1
Population: Participants using the Wisepill adherence monitor
Measure: Number; unit: participants
Arm/Group | SMS Reminders | No Reminders
Number analyzed (Participants) | 173 | 175
participants | 141 | 142
Statistical Analysis 1: Comparison: SMS Reminders vs No Reminders; Test type: Other — Pearson chi-square; p = 0.93, Chi-squared

3. Secondary Outcome: USD Per Month
Description: Cost estimates (including time and motion studies) and mathematical modeling estimate the cost-effectiveness of Wisepill plus SMS reminders per HIV case averted
Time Frame: two years
Population: Costs for study participants in the "SMS reminders" arm (data were not collected from participants in the "No Reminders" arm)
Measure: Number; unit: USD per month
Arm/Group | SMS Reminders | No Reminders
Number analyzed (Participants) | 173 | 0
USD per month
  Incremental cost per month in USD (Wisepill + SMS) | 12.64 |
  Incremental cost per month in USD (Wisepill + SMS; at scale) | 7.57 |
  Incremental cost per month in USD (SMS only) | 7.69 |
  Incremental cost per month in USD (SMS only; at scale) | 2.76 |

4. Other Pre Specified Outcome: Risk Perception
Description: Assess self-reported weekly HIV risk perception through an automated SMS survey
Time Frame: up to 2 years follow-up
Population: Number of participants by arm who reported perceived HIV risk during at least 1 week (among a subset of the participants responding to the SMS surveys)
Measure: Number; unit: participants
Arm/Group | SMS Reminders | No Reminders
Number analyzed (Participants) | 124 | 116
participants | 88 | 82
Statistical Analysis 1: Comparison: SMS Reminders vs No Reminders; Test type: Other — Pearson chi-square; p = 0.96, Chi-squared

5. Other Pre Specified Outcome: Adherence Measure Performance
Description: Tenofovir concentration in DBS compared to electronic adherence data from the prior 30 days for each participant.
Time Frame: up to 2 years follow-up
Population: Data reflect a 15% random sample.
Measure: Number; unit: Correlation coefficient
Arm/Group | SMS Reminders | No Reminders
Number analyzed (Participants) | 99 | 87
Correlation coefficient | 0.56 | 0.66

6. Other Pre Specified Outcome: Pregnancy Outcomes
Description: Descriptive measures of infants exposed to PrEP during gestation
Time Frame: 6 months post-partum or end of the study
Population: Number of pregnancies by arm
Measure: Count of Participants; unit: Participants
Arm/Group | SMS Reminders | No Reminders
Number analyzed (Participants) | 50 | 63
Participants
  live birth | 32 | 46
  pregnancy loss | 15 | 16
  ectopic | 2 | 0
  unknown | 1 | 1

ADVERSE EVENTS:
Time Frame: We attempted to follow all participants for 24 months.
Arm/Group | SMS Reminders | No Reminders
All-Cause Mortality (participants affected / at risk) | 1/173 | 0/175
Serious Adverse Events (participants affected / at risk) | 0/173 | 0/174
Other Adverse Events (participants affected / at risk) | 5/173 | 5/174
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SMS Reminders (N=173) | No Reminders (N=174)
Social harm (Social circumstances) | 5 | 5 — There were five social harms per study arm that were probably or definitely related to study participation, and consisted of verbal or physical abuse with a sexual partner.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-09-25): https://cdn.clinicaltrials.gov/large-docs/67/NCT02915367/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-04): https://cdn.clinicaltrials.gov/large-docs/67/NCT02915367/SAP_001.pdf